CLINICAL TRIAL: NCT02191163
Title: A 17 Week, Randomised, Double-blind, Placebo Controlled Cross-over Trial to Evaluate the Efficacy of Antistax® Film Coated Tablets (Extr. Vitis Vinifera Siccum), 360 mg/Day p.o. in Improving Microcirculation of the Skin in the Leg of Male and Female Patients Suffering From Chronic Venous Insufficiency
Brief Title: Efficacy of Antistax® in Improving Microcirculation of the Skin in the Leg in Patients Suffering From Chronic Venous Insufficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1138.3
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Venous Insufficiency
MeSH Terms: conditions — Venous Insufficiency | interventions — Antistax

ARMS (2):
- Antistax® (Experimental): 1 x 360 mg for 42 days
  Interventions: Drug: Antistax®
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Antistax®
  Arms: Antistax®
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to determine the efficacy and safety of Antistax® film coated tablets in improving microcirculation of the skin in the leg of patients with chronic venous insufficiency (CVI)

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* >= 18 years of age
* CVI I or CVI II (without expanded trophic disturbances)
* Willing and able to give written informed consent in accordance to Good Clinical Practice and local legislation prior to participation in the study

Exclusion Criteria:

Concomitant disease(s) exclusion criteria:

* Decompensated cardiac insufficiency
* Edema not due to venous disease of the legs (e.g. latent cardiac insufficiency, renal insufficiency, lymph edema, etc)
* Peripheral arterial disease (ankle/arm pressure index < 0.9)
* Current acute phlebitis or thrombosis
* Renal insufficiency (Serum creatinine > 1.5 mg/dl)
* Liver disease (SGPT (ALAT) > 3x upper limit of normal)
* Other diseases: insulin-dependent diabetes mellitus, neuropathies, hyper- or hypocalcaemia, malignancies
* Anamnestic indications of diabetic microangiopathy or polyneuropathy
* Drug and/or alcohol abuse
* Pregnant or nursing women or inadequate birth control methods (this applies to females of childbearing potential only)
* Severe climacteric complaints or changes in, or initiation with post-menopausal hormone replacement therapy within the last 3 months
* Immobility
* Avalvulie
* Klippel-Trénaunay-Weber-Syndrome (Naevus varicosis osteohypertrophicus, Haemangiectasia hypertrophicans)
* State after pulmonary embolism
* Recognized hypersensitivity to the trial drug ingredients
* Current florid venous ulcus
* Clinical indication for a necessary, specific phlebologic acute treatment, e.g. compressive treatment, phlebectomy, etc.

Previous treatment(s) exclusion criteria:

* Treatment with venous drugs within the last 4 weeks
* Changes in, or initiation with, treatment with theophylline, diuretics, cardiac glycosides, ACE inhibitors or calcium antagonists within the last 8 days

Concomitant treatment/non-drug therapy exclusion criteria:

* Other venous drugs apart from the trial medication
* Compression bandages
* Venous surgery of the leg used for the fluxmetry
* Extensive use (i.e. on more than a total of 6 days during the entire trial) of laxatives which affect fluid or electrolyte balance
* Major surgery requiring full anesthesia

Other exclusion criteria:

* Previously studied under this protocol
* Participation in another clinical trial within the previous 90 days or during the present study
* Patients considered as mentally ill as well as unable to work or with limited working ability, or unable (or only partially able) to follow the spoken or written explanations concerning the trial
* Patients in a bad general health state according to the investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2002-04; Primary Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in the resting flux | Baseline, after 6 weeks of treatment
  measured in the frequency range 10-37 kHz on the skin of the inside lower leg using the Laser Doppler Fluxmetry

SECONDARY OUTCOMES:
Changes from baseline in the resting flux | Baseline, after 3 weeks of treatment
  measured in the frequency range 10-37 kHz
Changes in the resting flux | Baseline, after 3 and 6 weeks of treatment
  measured in the frequency range <10 kHz
Changes in the combined resting fluxes (<37 kHz) | Baseline, after 3 and 6 weeks of treatment
Changes in the transcutaneous oximetry (TcPO2) | Baseline, after 3 and 6 weeks of treatment
  measured on the inside lower leg of the more CVI-affected leg
Change from baseline in the calf circumference of the most affected leg | Baseline, after 3 and 6 weeks of treatment
Change from baseline in the ankle circumference of the most affected leg | Baseline, after 3 and 6 weeks of treatment
Change from baseline in the subjective symptoms of CVI measured by Visual Analogue Scales (VAS) | Baseline, after 3 and 6 weeks of treatment
Global efficacy assessment by patient on a 4-point verbal rating scale (VRS) | after 6 weeks of treatment
Global efficacy assessment by investigator on a 4-point VRS | after 6 weeks of treatment
Number of patients with adverse events | up to 16 weeks
Number of patients with clinically relevant changes in laboratory values | Baseline, up to 16 weeks
Number of patients with clinically significant changes in vital signs | Baseline, up to 16 weeks
Global tolerability assessment by investigator on a 4-point VRS | after 6 weeks of treatment
Global tolerability assessment by patient on a 4-point VRS | after 6 weeks of treatment

REFERENCES:
- [Derived] Martinez-Zapata MJ, Vernooij RW, Simancas-Racines D, Uriona Tuma SM, Stein AT, Moreno Carriles RMM, Vargas E, Bonfill Cosp X. Phlebotonics for venous insufficiency. Cochrane Database Syst Rev. 2020 Nov 3;11(11):CD003229. doi: 10.1002/14651858.CD003229.pub4. PMID 33141449